CLINICAL TRIAL: NCT02543788
Title: CHRONIC OPTIC NEUROPATHY IN MULTIPLE SCLEROSIS: DEMYELINATING AND/OR PRIMARY DEGENERATIVE PATHOPHYSIOLOGY?
Brief Title: CHRONIC OPTIC NEUROPATHY IN MULTIPLE SCLEROSIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Collaborators: Fondation pour la Recherche Médicale (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2014.850
Record Dates: First submitted 2014-06-25; First posted 2015-09-07 (Estimated); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Chronic Optic Neuropathy in Multiple Sclerosis
Keywords: optic neuritis; vision; quality of life; pathophysiology
MeSH Terms: conditions — Optic Neuritis | interventions — Visual Acuity; Visual Fields; Color Vision

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- patients (Other): patients with chronic optic neuropathy in multiple sclerosis
  Interventions: Procedure: • Neuro-Ophthalmological examination, Visual Acuity, Fundus, Visual Field, Color Vision, OCT, EDSS • NEI-VFQ 25 and the 10-item • VEPs, p-ERG and mf-ERG
- Controls (Other): healthy volunteers
  Interventions: Procedure: • Neuro-Ophthalmological examination, Visual Acuity, Fundus, Visual Field, Color Vision, OCT, EDSS • NEI-VFQ 25 and the 10-item • VEPs, p-ERG and mf-ERG

INTERVENTIONS:
Procedure: • Neuro-Ophthalmological examination, Visual Acuity, Fundus, Visual Field, Color Vision, OCT, EDSS • NEI-VFQ 25 and the 10-item • VEPs, p-ERG and mf-ERG

SUMMARY:
Patients with multiple sclerosis (MS) may show chronic signs of optic neuropathy (CON) that may follow acute optic neuritis (secondary form of CON, S-CON) or occur independently of any acute demyelinating lesion of the optic nerve (primary form of CON, P-CON). In both S-CON and P-CON, a long term progressive ganglion cell axonal loss occurs. This axonal damage could be secondary to retrograde atrophy of axons within plaques of demyelination or a primary progressive degeneration of ganglion cells, but the underlying physiopathology has not been fully questioned in the different profile types of CON.

In this project, investigators aim at understanding the pathophysiology of S-CON and P-CON, i.e. secondary to demyelination or primary degeneration, in patients complaining of persistent visual complaints. In a first cross sectional study, 30 MS patients with mild to moderate P-CPON or S-CON and 30 age-matched control subjects will perform an extensive neuro-ophthalmological assessment including clinical examination, visual evoked potentials (pattern and low contrast), electroretinogram (pattern and multifocal ERG), OCT (peripapillary and macular volume scan segmentation protocols) and MRI of the optic nerve. In these patients with mild to moderate CON, investigators aim at differentiating patients showing predominant demyelination from those showing pure or predominant axonal degeneration. Visual function assessment and degree of axonal degeneration will be compared and correlated in the two types of underlying pathophysiology and in the group of control subject. In a following longitudinal study, the patients will be re-assessed a year later in order to evaluate the progression of CON in both profile types. Our hypothesis would be that visual function and progression is worse in the degeneration group as compared to the demyelination group. This study should help to find reliable measures of the pathophysiology of CON and correlate it with the long-term visual prognostic of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for patients

  * All patients may have a clinically definite, laboratory-supported diagnosis of multiple sclerosis according to the Mac Donald criteria (2010).
  * All patients may present a chronic visual complaint.
  * All patients may present mild to moderate chronic optic neuropathy (cf infra)
  * All patients may not have recent acute optic neuritis (<2 years)
  * All patients will be informed about the design and purpose of the study, and all will give their informed, written consent to the protocol, which may have been approved by the local ethics committee.
  * Age: > 18
  * Able to understand the instructions
  * Having a health coverage
  * Able to sit down for 1 hour Diagnosis of mild to moderate chronic optic neuropathy

For the diagnosis of optic neuropathy, patients will have to meet 3 of the 6 next criteria:

1. Far Visual Acuity (ETDRS charts, 100% contrast) < 85 letters
2. Far Visual Acuity (ETDRS charts, 2.5% contrast) < 60 letters
3. Mean visual field defect on static perimetry> 2dB
4. Mean pRNFL in OCT < 80 µ.
5. Color vision score > 35
6. Disc pallor Diagnosis of mild to moderate optic neuropathy

   * Far Visual Acuity (ETDRS charts, 100% contrast) >70 letters Diagnosis of chronic optic neuropathy
   * Stable or worsening of visual acuity, visual field and/or RNFL in OCT, at 6 month of interval

     - Inclusion criteria for controls
   * Age > 18 years
   * Visual acuity score (ETDRS) > 85
   * Able to understand the instructions
   * Having a health coverage
   * Informed and consenting to give his written consent

Exclusion Criteria:

* Non inclusion criteria for patients.

  * Ophthalmological

    * Other ophthalmological disorder that could impair corrected visual acuity (Maculopathy, Retinopathy…)
    * Ocular instability in primary position of gaze
  * Neurological

    * Ongoing seizure
    * Severe handicap that does not allow sitting down position for 1 hour
  * General

    * Unstable medical state
    * Severe renal insufficiency
    * Allergy to gadolinium
    * Claustrophobia
    * Implanted electrical stimulator (pace maker)
    * Metallic prosthesis or orthesis, cochlear implants
    * Intraocular foreign material
  * Pregnancy (on questioning)
  * Tutelage or any legal protection measure
* Non inclusion criteria for controls

  * Any ophthalmological disorder that could impair corrected visual acuity
  * Any neurological disorder
  * MRI contraindication
  * Allergy to gadolinium
  * Severe renal insufficiency
  * Claustrophobia
  * Implanted electrical stimulator (pace maker)
  * Metallic prosthesis or orthesis, cochlear implants
  * Intraocular foreign material
  * Pregnancy (on questioning)
  * Tutelage or any legal protection measure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change from Day0 15' P100 VEP latency at one year | D0 and one year
  15' VEP latency may be the best outcome that allow differentiating patients from controls, and each of the sub-group of patients

SECONDARY OUTCOMES:
Change from Day0 100%, 2.5% and 1.25% ETDRS Visual Acuity at one year (composite measure) | D0 and one year
Change from Day0 Visual field macular threshold and corrected mean visual field deficit at one year (composite measure) | D0 and one year
change frome Day0 NEI-VFQ 25 composite score and 10-item score at one year (composite measure) | D0 and one year
Change from Day0 N75, P100, N135 VEP latency and amplitude; P50, N95 ERG latency and amplitude; p1 mERG latency and amplitude at one year (composite measure) | D0 and one year
Change from Day0 OCT peripapillary RNLF thickness and Ganglion cell layer average thickness on macular dense volume at one year (composite measure) | D0 and one year
MRI presence or absence of optic nerve inflammatory signs on diameter of the optic nerve | D0

CONTACTS AND LOCATIONS:
Overall Officials: Caroline TILIKETE, MD, Principal Investigator — Unité de Neuro-Ophtalmologie - Hôpital Neurologique - HOSPICES CIVILS DE LYON - France
Locations (1):
- Unité de Neuro-Ophtalmologie - Hôpital Neurologique - HOSPICES CIVILS DE LYON, France, BRON, France

REFERENCES:
- [Background] Physiopathologie de la Neuropathie Optique Chronique de la SEP " Lucie ABOUAF, François DURAND-DUBIEF, Sandra VUKUSIC, Alain VIGHETTO, Caroline TILIKETE. Communication orale aux 3e journée des Neurosciences de l'Hôpital Neurologique le jeudi 24 septembre 2015, Institut des Sciences Cognitives, Lyon.